CLINICAL TRIAL: NCT02279134
Title: A Phase II/III Study of Adjuvant Chemoradiotherapy, Radiotherapy After Surgery Versus Surgery Alone in Patients With Stage ⅡB-Ⅲ Esophageal Carcinoma
Brief Title: Phase II/III Study Compare Adjuvant Chemoradiotherapy, Radiotherapy and Surgery Alone for Esophageal Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zefen Xiao (Unknown)
Responsible Party: Sponsor-Investigator, Zefen Xiao, Chinese Academy of Medical Sciences, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-090/880
Record Dates: First submitted 2014-10-26; First posted 2014-10-30 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Esophageal Neoplasms; Esophageal Cancer
Keywords: StageⅡB-Ⅲ esophageal cancer; adjuvant radiotherapy; adjuvant chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Cisplatin; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Surgery alone (No Intervention): No adjuvant treatment after radical resection is developed in this arm
- Adjuvant Chemoradiation (Experimental): Adjuvant chemoradiation after radical resection is developed in this arm
  Interventions: Radiation: Adjuvant Chemoradiation; Drug: Paclitaxel; Drug: Cisplatin or Nedaplatin
- Adjuvant Radiation (Active Comparator): Adjuvant radiation after radical resection is developed in this arm
  Interventions: Radiation: Adjuvant Radiation

INTERVENTIONS:
Radiation: Adjuvant Chemoradiation — Patients receive Paclitaxel 135-150mg/m2 (D1 and D29) and Cisplatin or Nedaplatin 50-75mg/m2 (D1 and D29) every 4 weeks, concurrent with radiotherapy. Prophylactic polyethylene glycol recombinant human G-CSF is administered 48 hours after chemotherapy. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Arms: Adjuvant Chemoradiation
Radiation: Adjuvant Radiation — Patients undergo radiotherapy once daily 5 days a week for an average of 5.5 weeks within 12 weeks after surgery in the absence of disease progression or unacceptable toxicity.
  Arms: Adjuvant Radiation
Drug: Paclitaxel — 135-150mg/m2 (D1 and D29)
  Arms: Adjuvant Chemoradiation
Drug: Cisplatin or Nedaplatin — 50-75mg/m2 (D1 and D29)
  Arms: Adjuvant Chemoradiation

SUMMARY:
This phase III trial is studying how well the combination of chemoradiation or radiation works in resected locally advanced cancer of the esophagus or gastroesophageal junction.

DETAILED DESCRIPTION:
Although preoperative chemoradiation therapy followed by surgery is the most common approach for patients with resectable esophageal cancer, considerable number of esophageal cancer patients received operation as the first treatment modality. Accordingly, postoperative treatments have always been playing an important role because of the poor survival rates of the patients in stage ⅡB[UICC 7th edition] -Ⅲ[UICC 7th edition] who have been treated with resection alone. The existing data shows that the 5-yeal survival rate of stageⅡB-Ⅲ of thoracic esophageal squamous cell carcinoma(TESCC) after surgery is merely about 28.4% ,and locoregional lymph nodes metastases is responsible for the main cause of failure. While we have proved the value of prophylactic radiation therapy after radical esophagectomy for esophageal carcinoma with positive lymph node metastases and stage Ⅲ disease (UICC 6th edition) under the conventional 2-dimensional radiotherapy methods in subset analysis of prospective randomized clinical trial. For patients with positive lymph nodes, 5 year survival after surgery alone was 28.4%, median overall survival was 24 months, recurrence patterns were 34.6% in mediastinal lymph nodes，13.3% in supraclavicular lymph nodes，10% in abdominal lymph nodes. Distant metastases occurred in 21% patients. Adjuvant radiotherapy significantly reduced the recurrence in mediastinal lymph nodes(13.4%), supraclavicular lymph nodes (6.1%). However distant metastases rate increased to 30.7%. Chemotherapy may be vital for these patients. Chen reported that 5 year overall survival rates for the chemoradiotherapy group and radiotherapy group were 47.4% and 38.6% (P=0.03). Based on our studies, treatment failure occurred in 8% patients because of celiac metastases. Small radiation field by omitting celiac drainage region may ensure patients to accept 2 cycles of concurrent chemotherapy for lower toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. KPS≥70
2. Diagnosis of stage ⅡB or Ⅲ thoracic esophageal cancer
3. Complete resection
4. Adequate organ function:

Hematopoietic Absolute granulocyte count at least 1,500/mm^3 Platelet count at least 150,000/mm^3 Hemoglobin at least 10 g/dL Hepatic Not specified Renal Creatinine no greater than 1.5 mg/dL AND/OR Creatinine clearance at least 65 mL/min Calcium no greater than 11 mg/dL Cardiovascular No uncontrolled heart disease No uncontrolled hypertension

Exclusion Criteria:

1. Uncontrolled diabetes
2. Interval between surgery and adjuvant therapy more than 3 months
3. Sign of recurrence on CT scan or ultrasound or PET-CT No palpable subclavicular lymph nodes or involvement after cytology needle aspiration No lymph nodes greater than 1 cm on CT scan
4. With Weight loss greater than 10% from baseline
5. With other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
6. Be pregnant

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | up to 3 years
  From the date of randomization to the date of first failure or last follow-up

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years
  From the date of randomization to the date of death or last follow-up

OTHER OUTCOMES:
Adverse events | up to 5 years
  From the date of randomization to the date of death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Zefen Xiao, MD, Principal Investigator — Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Science
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Xiao ZF, Yang ZY, Liang J, Miao YJ, Wang M, Yin WB, Gu XZ, Zhang DC, Zhang RG, Wang LJ. Value of radiotherapy after radical surgery for esophageal carcinoma: a report of 495 patients. Ann Thorac Surg. 2003 Feb;75(2):331-6. doi: 10.1016/s0003-4975(02)04401-6. PMID 12607634
- [Background] Xiao ZF, Yang ZY, Miao YJ, Wang LH, Yin WB, Gu XZ, Zhang DC, Sun KL, Chen GY, He J. Influence of number of metastatic lymph nodes on survival of curative resected thoracic esophageal cancer patients and value of radiotherapy: report of 549 cases. Int J Radiat Oncol Biol Phys. 2005 May 1;62(1):82-90. doi: 10.1016/j.ijrobp.2004.08.046. PMID 15850906
- [Background] Chen J, Zhu J, Pan J, Zhu K, Zheng X, Chen M, Wang J, Liao Z. Postoperative radiotherapy improved survival of poor prognostic squamous cell carcinoma esophagus. Ann Thorac Surg. 2010 Aug;90(2):435-42. doi: 10.1016/j.athoracsur.2010.04.002. PMID 20667325
- [Background] Mariette C, Balon JM, Piessen G, Fabre S, Van Seuningen I, Triboulet JP. Pattern of recurrence following complete resection of esophageal carcinoma and factors predictive of recurrent disease. Cancer. 2003 Apr 1;97(7):1616-23. doi: 10.1002/cncr.11228. PMID 12655517
- [Background] Teniere P, Hay JM, Fingerhut A, Fagniez PL. Postoperative radiation therapy does not increase survival after curative resection for squamous cell carcinoma of the middle and lower esophagus as shown by a multicenter controlled trial. French University Association for Surgical Research. Surg Gynecol Obstet. 1991 Aug;173(2):123-30. PMID 1925862
- [Background] Fok M, Sham JS, Choy D, Cheng SW, Wong J. Postoperative radiotherapy for carcinoma of the esophagus: a prospective, randomized controlled study. Surgery. 1993 Feb;113(2):138-47. PMID 8430362
- [Background] Zieren HU, Muller JM, Jacobi CA, Pichlmaier H, Muller RP, Staar S. Adjuvant postoperative radiation therapy after curative resection of squamous cell carcinoma of the thoracic esophagus: a prospective randomized study. World J Surg. 1995 May-Jun;19(3):444-9. doi: 10.1007/BF00299187. PMID 7639004
- [Derived] Ni W, Xiao Z, Zhou Z, Chen D, Feng Q, Liang J, Lv J. Severe radiation-induced lymphopenia during postoperative radiotherapy or chemoradiotherapy has poor prognosis in patients with stage IIB-III after radical esophagectomy: A post hoc analysis of a randomized controlled trial. Front Oncol. 2022 Sep 8;12:936684. doi: 10.3389/fonc.2022.936684. eCollection 2022. PMID 36158699
- [Derived] Ni W, Yu S, Zhang W, Xiao Z, Zhou Z, Chen D, Feng Q, Liang J, Lv J, Gao S, Mao Y, Xue Q, Sun K, Liu X, Fang D, Li J, Wang D. A phase-II/III randomized controlled trial of adjuvant radiotherapy or concurrent chemoradiotherapy after surgery versus surgery alone in patients with stage-IIB/III esophageal squamous cell carcinoma. BMC Cancer. 2020 Feb 18;20(1):130. doi: 10.1186/s12885-020-6592-2. PMID 32070309
- See also: It is a national center for cancer research and treatment. It is one of the clinical trial bases approved by the Food and Drug Administration of State (SFDA) — http://www.cicams.ac.cn